CLINICAL TRIAL: NCT05993637
Title: A Comparison of the Effects of High Tibial Osteotomy and Unicompartmental Knee Arthroplasty Surgeries on Proprioception Applied to Individuals With Medial Gonarthrosis
Brief Title: Comparison of Proprioception for HTO (High Tibial Osteotomy) and UKA (Unicompartmantal Knee Arthroplasty)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: F-473945936
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
Keywords: Gonarthrosis; High Tibial Osteotomy; Unicompartmantal Knee Arthrodesis; Proprioception
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Tibial Osteotomy: patients who were diagnosed with medial gonarthrosis and underwent HTO surgery
  Interventions: Other: Examination of propriception
- Unicompartmantal Knee Arthroplasty: patients who were diagnosed with medial gonarthrosis and underwent UKA surgery
  Interventions: Other: Examination of propriception

INTERVENTIONS:
Other: Examination of propriception — application of the tests used in proprioception assessment to patients by a physiotherapist

SUMMARY:
Osteoarthritis of the knee (KOA), a common degenerative joint disease, affects a significant part of the world's population. Although it can hold all the compartments in the knee joint, isolated medial compartment involvement has been reported in about 85% of individuals diagnosed with KOA.

In the management of degenerative medial gonarthrosis; symptomatic relief and provide orthopaedic surgeons with the aim to slow down the progression of Total Knee Arthroplasty (TKA) unikompartmental knee arthroplasty (UKA) and high tibial osteotomy (HTO) is used. In recent years, HTO and UKA have been preferred more frequently among these surgical methods due to a number of advantages they provide for patients.

As a result of the orthopedic surgeries performed, interventions are made on bone and joint structures and problems may occur in the proprioceptive inputs provided by the body. In UKA, a new joint structure is created by changing the bone structure and removing the tibial plateau, while in HTO, the existing bone structure is preserved and a positional change is created. Thus, while it is expected that the proprioceptive response to be different between the two surgeries, no studies have been found in the literature on this issue. Accordingly, the purpose of this study is to compare the effects of HTO and UKA surgeries applied to individuals diagnosed with medial gonarthrosis on the proprioception of patients and to examine the effects of HTO and UKA surgeries on patients diagnosed with medial gonarthrosis.

H0: There is no difference between the surgical methods applied when the proprioception of patients with HTO and UKA surgeries planned for individuals with medial gonarthrosis is considered.

H1: There is a difference between the surgical methods applied when the proprioception of patients with HTO and UKA surgeries planned for individuals with medial gonarthrosis are considered.

DETAILED DESCRIPTION:
Volunteer participants who have been diagnosed with medial gonarthrosis and have varus deformity and have undergone surgery will be included. The surgical groups will be divided into two categories: HTO and UKA. Evaluations of the participants in terms of proprioception will be made. A voluntary consent form will be obtained from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery at the age of 50-65
* Performing unilateral UKA or HTO surgery
* Moderate medial knee arthrosis on pre-op X-ray
* Presence of mild varus deformity in the pre-op period
* Should be BMI<30

Exclusion Criteria:

* Regular exercise at least 3 days a week, 150 minutes, moderate intensity
* Having undergone revision surgery
* The presence of any other orthopedic problems/problems and surgery
* Concomitant of a common rheumatological disease
* Presence of neurological problems/problems
* Having visual and auditory problems at a level that prevents communication

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with medial gonarthrosis and undergone surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Romberg Test | Day 1
  The patient is asked to stand in an upright position with his feet open at shoulder level and his arms free at the sides. The patient, who does not receive any support, is asked to stand first with his eyes open and then with his eyes closed. While the patient is standing still, the time until the moment when his balance is disturbed is recorded.

SECONDARY OUTCOMES:
Knee Society Score | Day 1
  The system is divided into a knee score, which assesses only the knee joint itself, and functional scores, which assesses the patient's ability to walk and climb stairs. As a result of the dual rating system, the problem of decreasing knee scores associated with patient weakness is eliminated.
WOMAC | Day 1
  It is a scale that evaluates the disability associated with these conditions in hip and/or knee osteoarthritis. It consists of three parts: pain, stiffness and physical function. It contains a total of 24 substances.
Single Leg Stance Test | Day 1
  It is used to evaluate static posture and balance control. The patient should stand unaided on one leg from the moment when the other foot leaves the floor until the time when the foot touches the floor again or the arms leave the hips.
5-times Sit to Stand Test | Day 1
  It is used to assess the functional strength of the lower extremities, transitional movements, balance and the risk of falls. Participants are evaluated by sitting on a back-supported chair five times and holding it for a while while getting up.
change from baseline Gait Analyzer for walking speed at 8 weeks (m/sec) | Day 1
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step duration, step length, cadence and symmetry.
change from baseline Gait Analyzer for step time at 8 weeks (sec) | Day 1
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step duration, step length, cadence and symmetry.
change from baseline Gait Analyzer for step lenght at 8 weeks (m) | Day 1
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step duration, step length, cadence and symmetry.
change from baseline Gait Analyzer for cadance at 8 weeks (step/min) | Day 1
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step duration, step length, cadence and symmetry.
change from baseline Gait Analyzer for symmetry at 8 weeks (%) | Day 1
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step duration, step length, cadence and symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan Karagoz, Prof., Study Director — Istanbul University - Cerrahpasa

REFERENCES:
- [Background] Willis-Owen CA, Brust K, Alsop H, Miraldo M, Cobb JP. Unicondylar knee arthroplasty in the UK National Health Service: an analysis of candidacy, outcome and cost efficacy. Knee. 2009 Dec;16(6):473-8. doi: 10.1016/j.knee.2009.04.006. Epub 2009 May 22. PMID 19464898
- [Background] Johal S, Nakano N, Baxter M, Hujazi I, Pandit H, Khanduja V. Unicompartmental Knee Arthroplasty: The Past, Current Controversies, and Future Perspectives. J Knee Surg. 2018 Nov;31(10):992-998. doi: 10.1055/s-0038-1625961. Epub 2018 Mar 7. PMID 29514367
- [Background] Cao Z, Mai X, Wang J, Feng E, Huang Y. Unicompartmental Knee Arthroplasty vs High Tibial Osteotomy for Knee Osteoarthritis: A Systematic Review and Meta-Analysis. J Arthroplasty. 2018 Mar;33(3):952-959. doi: 10.1016/j.arth.2017.10.025. Epub 2017 Dec 2. PMID 29203354
- [Background] He M, Zhong X, Li Z, Shen K, Zeng W. Progress in the treatment of knee osteoarthritis with high tibial osteotomy: a systematic review. Syst Rev. 2021 Feb 14;10(1):56. doi: 10.1186/s13643-021-01601-z. PMID 33583421
- [Background] Santoso MB, Wu L. Unicompartmental knee arthroplasty, is it superior to high tibial osteotomy in treating unicompartmental osteoarthritis? A meta-analysis and systemic review. J Orthop Surg Res. 2017 Mar 28;12(1):50. doi: 10.1186/s13018-017-0552-9. PMID 28351371
- [Background] Ghai S, Driller M, Ghai I. Effects of joint stabilizers on proprioception and stability: A systematic review and meta-analysis. Phys Ther Sport. 2017 May;25:65-75. doi: 10.1016/j.ptsp.2016.05.006. Epub 2016 May 18. PMID 28262354